CLINICAL TRIAL: NCT06300385
Title: Effect of Electromyostimulation and Strengthening Exercises on Pain, Fatigue and Physical Performance in Motocross Athletes
Brief Title: Effect of EMS and Strengthening Exercises on Pain, Fatigue and Physical Performance in Motocross Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Furkan Çakır, Principal Investigator, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulBUFC5
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Sports Injury
Keywords: sports; electromyostimulation; exercise; pain; fatigue; strength
MeSH Terms: conditions — Athletic Injuries; Motor Activity; Pain; Fatigue

STUDY DESIGN:
Intervention Model Description: 2 parallel groups randomized controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): These participants will receive electromyostimulation simultaneously with strengthening exercise.
  Interventions: Device: Electromyostimulation; Other: Strengthening exercises
- Sham control (Sham Comparator): These participants will receive sham electromyostimulation (current turned off) simultaneously with strengthening exercise.
  Interventions: Other: Strengthening exercises

INTERVENTIONS:
Device: Electromyostimulation — Electromyostimulation (EMS), a low-frequency current, will be used for electrical stimulation of the wrist flexor muscle group. Stimulation frequency will be applied as 25 Hertz. Care will be taken to ensure that the current intensity does not cause pain in the patient. The size of the EMS electrodes is 2 cm2 and they will be placed in the form of 4 electrodes on the wrist flexor muscles (inner wrist area) with a distance of 1 cm between them. Each strengthening session will be 15 minutes for 6 weeks, 3 days a week, for a total of 18 sessions. EMS application will be carried out together with strengthening exercises. Laica MD6078 branded device belonging to the researchers will be used.
  Arms: Experimental
Other: Strengthening exercises — All participants will do resistance exercises for strengthening, 3 sessions per week for 6 weeks. Each movement will be performed in 3 sets and 12 repetitions according to the planned intensity. Wrist curl, reverse wrist curl movements (with 10kg dumbbells) and power web flex grip movements will be applied simultaneously with EMS application. The program will last 15 minutes in total.

SUMMARY:
Motocross, a popular sport, involves riding motorized vehicles on rugged tracks with obstacles. It's physically demanding, with high speeds and a risk of accidents. Grip strength is crucial, especially in the arms and forearms, which are prone to injury. Physiotherapy often employs strength exercises, including electromyostimulation. However, there's little research on their effectiveness for motocross athletes. This study aims to compare electromyostimulation combined with strength training versus strength training alone in relieving pain, fatigue, and improving strength in motocross athletes.

DETAILED DESCRIPTION:
Motocross is a popular sport in which participants ride a two-wheeled, motorized vehicle around a 2 km rugged track with natural or man-made obstacles. Participants race at high speeds and it is considered a strenuous sport with a high accident rate. Motocross racers grip the handlebars of their bikes with both hands throughout the race, which lasts between 18 and 26 minutes. Therefore, it is a sports branch where control is concentrated on the arms and upper extremities. It has been reported that the most frequently injured and painful area is the forearm. Therefore, good and strong upper extremity and forearm control is important for the prevention of injuries or subsequent recovery processes.

It is known that strengthening exercise programs are used in physiotherapy practices to improve strength and stabilization parameters. The use of electromyostimulation applications for strengthening in different populations is also becoming widespread.

There are no studies demonstrating the effectiveness of strengthening and electromyostimulation applications on pain, fatigue and strength parameters in motocross athletes.

The aim of this study is to compare the effectiveness of electromyostimulation application applied simultaneously with a strengthening exercise program on pain, fatigue and strength, with strengthening exercises performed with sham application (electric current turned off).

ELIGIBILITY:
Inclusion Criteria:

* Having at least 5 years of professional motocross training experience
* Being between 18 and 30 years old
* Volunteering to participate in the study

Exclusion Criteria:

* To be absent from the 6-week EMS and strengthening program for more than 2 consecutive sessions
* Having suffered any injury that prevents you from training in the last 6 months
* Being receiving a physiotherapy program other than the protocol to be used in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 6 week
  Pain assessment: Pain scores of patients will be recorded using 0-100 mm Visual Analog Scale (VAS) to grade pain. For VAS; A measured horizontal line will be created, and definitions such as 'no symptoms' and 'severe symptoms' will be written at both ends. The participant will be instructed to mark a point on the line appropriate to the severity of the symptom. Wrist pain values in the resting position will be recorded before and after the 6-week program.
Strength measurement | 6 week
  Lafayette Dynamometer: Lafayette Manual Muscle Testing device will be used to evaluate muscle strength. While the measurements are being made, the device will be kept stationary and the resistance given by the participant will be measured in Newtons. Measurements will be made in the sitting position for wrist flexion/extension and forearm flexion, and total muscle strength will be recorded.
Fatigue assessment | 6 week
  Fatigue Severity Scale: The fatigue level of the participants will be evaluated with the Fatigue Severity Scale. It is a survey with 9 questions and 8-point Likert form.A high score means a high level of fatigue.
Grip strength assessment | 6 week
  Jamar Hand Grip Dynamometer will be used to evaluate hand grip and finger flexor muscle strength. The participant will sit upright during the assessment. Elbow and knee angle will be 90 degrees. A full force grip will be required with the wrist in the neural position. The measurement will be performed 3 times with an interval of 10 seconds. Increasing values will indicate higher strength. Measurement results will be recorded in kilograms and pounds.

CONTACTS AND LOCATIONS:
Overall Officials: Hulya Sisli, PhD, Study Director — Istanbul Bilgi University
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No